CLINICAL TRIAL: NCT00175240
Title: Enhancing the Use of Secondary Prevention Strategies in Patients With Coronary Artery Disease (The ESP-CAD Study)
Brief Title: Enhancing the Secondary Prevention of Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Alberta Heritage Foundation for Medical Research (Other); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UofA M2022
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Disease; Ischemic Heart Disease
Keywords: Coronary disease; quality improvement; knowledge translation
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia

INTERVENTIONS:
Behavioral: Evidence summaries endorsed by local opinion leaders

SUMMARY:
People with coronary artery disease can reduce their chance of having a heart attack by making healthy lifestyle choices (diet, exercise, quitting smoking,etc.). There are also many medications that have been proven to reduce the risk of heart attacks and may even help people live longer. This study will look at different ways of improving the use of these beneficial medications to enhance the quality of care for people with this condition.

DETAILED DESCRIPTION:
BACKGROUND: Despite the abundant evidence base for secondary prevention, practice audits consistently demonstrate substantial "care gaps" between this evidence and clinical reality such that many patients with Coronary Artery Disease (CAD) are not offered all possible therapies for the prevention of myocardial infarction or death. For example, even after an acute myocardial infarction, almost one fifth of patients continue to smoke; over half with hypertension or hyperlipidemia have poorly controlled pressure or lipid levels; and proven therapies such as statins, ACE inhibitors, beta-blockers and antiplatelet agents are under-prescribed.

Multiple barriers are often responsible for the lack of implementation of proven efficacious therapies and traditional means of educating practitioners (journal articles, CME, conferences, etc) are usually ineffective in altering practice. Clearly novel interventions to improve the quality of prescribing are needed. Local opinion leaders are trusted by their peers to evaluate medical innovations and thus influence practice patterns within their community. Few controlled studies, however, have evaluated their effect on changing prescribing practices for common conditions such as CAD.

HYPOTHESIS: This trial will test 2 quality improvement interventions. The principle hypothesis is: does a one-page evidence summary endorsed by local opinion leaders increase the provision of secondary prevention therapies in patients with CAD compared to usual care? The secondary hypotheses are: does the same intervention but without local opinion leader endorsement improve the provision of secondary prevention strategies in patients with CAD compared to usual care? Does local opinion leader endorsement increase the effectiveness of the quality improvement intervention?

ELIGIBILITY:
Inclusion Criteria:

* Alberta residents who undergo a cardiac catheterization and are diagnosed with coronary artery disease (> or equal to 50% stenosis in at least one vessel).

Exclusion Criteria:

* no fasting lipid panel within the previous 6 weeks
* on a statin at maximal dose
* on a statin/lipid lowering drug and LDL-C is 2.5 mmol/L or less (prior to Sept 2006) and LDL-C is 2.0 mmol/L or less (after Sept 2006)
* not on a statin and LDL-C is 1.8 mmol/L or less
* acute myocardial infarction or cardiogenic shock
* require emergency bypass surgery following catheterization
* contraindication to statins (e.g. cirrhosis, inflammatory muscle disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2005-03; Primary Completion 2011-08 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Composite measure representing improvement in cholesterol-related secondary prevention consisting of (1) provision of a statin sample (2) provision of a statin prescription or (3) dosage increase of a statin within the first 6 months post-angiogram.

SECONDARY OUTCOMES:
Provision of other proven efficacious medications for coronary artery disease by 6 months including ACE inhibitors, beta-blockers and antiplatelet agents.
Changes in the provision of other lipid lowering medications.
Smoking rates - receipt of smoking cessation advice/nicotine replacement products/bupropion.
Repeat fasting lipid panel within 6 months post-angiogram.
Proportion of patients achieving target LDL-C of 2.0mmol/l or less.
Clinical events including myocardial infarction, stroke, admissions for coronary artery disease, total hospitalizations and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Finlay McAlister, MD,MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital; Royal Alexandra Hospital, Foothills Medical Centre (Calgary), Edmonton, Alberta, Canada

REFERENCES:
- [Background] McAlister FA, Fradette M, Graham M, Majumdar SR, Ghali WA, Williams R, Tsuyuki RT, McMeekin J, Grimshaw J, Knudtson ML. A randomized trial to assess the impact of opinion leader endorsed evidence summaries on the use of secondary prevention strategies in patients with coronary artery disease: the ESP-CAD trial protocol [NCT00175240]. Implement Sci. 2006 May 6;1:11. doi: 10.1186/1748-5908-1-11. PMID 16722548
- [Result] McAlister FA, Fradette M, Majumdar SR, Williams R, Graham M, McMeekin J, Ghali WA, Tsuyuki RT, Knudtson ML, Grimshaw J. The Enhancing Secondary Prevention in Coronary Artery Disease trial. CMAJ. 2009 Dec 8;181(12):897-904. doi: 10.1503/cmaj.090917. Epub 2009 Nov 23. PMID 19933787
- [Result] McAlister FA, Majumdar SR, Lin M, Bakal J, Fradette M, Anderson T. Cholesterol end points predict outcome in patients with coronary disease: quality improvement metrics from the enhancing secondary prevention in coronary artery disease (ESP-CAD) trial. Can J Cardiol. 2014 Dec;30(12):1627-32. doi: 10.1016/j.cjca.2014.07.008. Epub 2014 Jul 16. PMID 25307535